CLINICAL TRIAL: NCT00098319
Title: Oral Cleft Prevention Trial in Brazil
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NICHD Global Network for Women's and Children's Health (Network)
Collaborators: Global Network for Women's and Children's Health Research (Other); Bill and Melinda Gates Foundation (Other); National Institute of Dental and Craniofacial Research (NIDCR) (NIH); Fogarty International Center of the National Institute of Health (NIH); National Center for Complementary and Integrative Health (NCCIH) (NIH); National Cancer Institute (NCI) (NIH); RTI International (Other); University of Iowa (Other); Hospital de Reabilitação de Anomalias Craniofaciais (HRAC) - Brazil (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GN 04 Aim III
Record Dates: First submitted 2004-12-06; First posted 2004-12-07 (Estimated); Last update posted 2013-12-17 (Estimated); Status verified 2013-12

CONDITIONS: Cleft Lip; Cleft Palate
Keywords: Cleft palate; Cleft lip; Folic acid; Global Network; Maternal and child health; International; Women's health; Brazil; Brasil; Latin America; ECLAMC; Congenital defects; Pregnancy
MeSH Terms: conditions — Cleft Lip; Cleft Palate; Congenital Abnormalities | interventions — Folic Acid

INTERVENTIONS:
Drug: Folic acid (0.4mg vs. 4.0mg)

SUMMARY:
Cleft lip and palate are a significant component of morbid human birth defects in the developing world. By supplementing a high-risk group of women with folic acid (4.0 mg versus 0.4 mg) from preconception and continuing throughout the first 3 months of pregnancy in the state of Sao Paulo, Brazil, this study aims to reduce the recurrence of cleft lip and palate.

DETAILED DESCRIPTION:
Craniofacial anomalies and cleft lip with or without cleft palate (CL/P) are a model for the impact of birth defects on fetal and neonatal health directly and maternal health indirectly. Craniofacial anomalies comprise a significant component of morbid human birth defects. The primary hypothesis is that folic acid supplementation of 4mg/day at preconception and during the first three months of pregnancy will decrease the recurrence of nonsyndromic cleft lip with or without clef palate (NSCL/P) in a high-risk group of women when compared to women taking 0.4 mg per day of folic acid. The total sample will include 2,000 women (that either have NSCL/P or that have at least one child with NSCL/P) randomly assigned to the 4 mg versus the 0.4 mg folic acid study groups. The study will also compare the recurrence rates of NSCL/P in the total sample of subjects as well as the two study groups (4mg, 0.4 mg) to that of a historical control group.

The primary outcome assessed is the rate of recurrences of NSCL/P in offspring of the trial mothers in each of the two study groups. Secondary outcomes include recurrence of NSCL/P compared to a historical control group; serum and red cell folate levels; severity of NSCL/P in offspring of trial mothers; twinning rate; miscarriage rate; preeclampsia; rates of other birth defects; birth weight; and gestational age. The sample size was based on historic tables of birth rates and the rates of cleft occurrences. The study hypothesizes that a total of 2000 subjects will be enrolled during a 2.5 year period; a dropout rate of 10%; birth rate for group A (women with NSCL/P) of 10% and a rate of 12% for group B (women with at least one child with NSCL/P); risk of cleft for group A is 7% and for group B is 4%; one-sided test with continuity correction.

ELIGIBILITY:
Inclusion Criteria:

* All women must reside in the state where the clinic is located.
* Women with NSCL/P who attend the craniofacial clinics, who are 16 to 45 years of age (after age 45 fecundity decreases substantially)who attend the craniofacial clinic for their care.
* Women (ages 16 to 45 years of age) who have at least one natural child of any age with NSCL/P who receives care at the participating craniofacial clinics.

Exclusion Criteria:

* Cases resulting from consanguineous couples (first, second, and third degree, i.e., first cousins or closer).
* Couples where at least one of the two is definitely sterilized.
* Women on anti-epileptic drugs.
* Women who are pregnant.
* Women who are planning to move outside of the state where the clinic is located within the next year.
* Women who are planning to move outside of Sao Paulo state within the next year.
* Women who have B12 deficiency (B12 level is below 174 pg/ml or 134.328 pmol/L).
* Women who have an allergy to folic acid.

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 2200 (Estimated)
Dates: Start 2004-01; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Recurrence of nonsyndromic cleft lip with or without cleft palate (NSCL/P) in offspring of trial mothers

SECONDARY OUTCOMES:
Recurrence of NSCL/P compared to a historical control group; Overall and high versus low dose
Serum and red cell folate levels
Severity of NSCL/P in offspring of trial mothers
Twinning rate
Miscarriage rate
Preeclampsia
Rates of other birth defects
Birth weight
Gestational age

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Murray, M.D., Principal Investigator — University of Iowa
Locations (3):
- Brazil (3):
  - Hospital de Reabilitação de Anomalias Craniofaciais (HRAC), Bauru, São Paulo
  - Hospital de Clinicas de Porto Alegre (HCPA), Porto Alegre
  - Hospital Santo Antonio-Centrinho: Obras Sociais Irma Dulce, Salvador

REFERENCES:
- See also: Global Network for Women's and Children's Health Research — http://gn.rti.org/
- See also: RTI International — http://www.rti.org/